CLINICAL TRIAL: NCT01235689
Title: An Open-Label, Multicenter, Efficacy and Safety Study to Evaluate Two Treatment Algorithms in Subjects With Moderate to Severe Crohn's Disease
Brief Title: Efficacy and Safety of Two Treatment Algorithms in Adults With Moderate to Severe Crohn's Disease
Acronym: CALM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M11-271; 2010-020137-10 (EudraCT Number)
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab; Prednisone; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tight Control Management (Experimental): Participants randomized to receive management of disease activity using criteria based on Crohn's Disease Activity Index (CDAI), high sensitivity C-reactive protein (hs-CRP), fecal calprotectin, and corticosteroid use.
  Participants received customized therapy that could include prednisone, adalimumab, and azathioprine. Participants who randomized at Week 9 meeting success criteria started with no therapy; participants who randomized prior to Week 9 or who randomized at Week 9 but did not meet the success criteria began treatment with adalimumab.
  Therapy was escalated according to pre-specified tight control criteria: At Key Visit 1 the success criteria were CDAI < 150, hs-CRP, < 5 mg/L, fecal calprotectin < 250 μg/g, and absence of prednisone use. At Key Visits 3, 4, and 5 (every 12 weeks after Key visit 1), the criteria were CDAI < 150, hs-CRP < 5 mg/L, fecal calprotectin < 250 μg/g, and absence of prednisone during the preceding week.
  Interventions: Biological: Adalimumab; Drug: Prednisone; Drug: Azathioprine
- Clinically Driven Management (Active Comparator): Participants randomized to receive management of disease activity using criteria based on Crohn's Disease Activity Index (CDAI) and corticosteroid use.
  Participants received customized therapy that could include prednisone, adalimumab, and azathioprine.
  Participants who randomized at Week 9 meeting success criteria started with no therapy; participants who randomized prior to Week 9 or who randomized at Week 9 but did not meet the success criteria began treatment with adalimumab.
  Therapy was escalated according to pre-specified failure criteria using less stringent criteria:
  At Key Visit 1 the criteria for management of disease activity were a CDAI decrease ≥ 70 (CR-70) compared to Baseline or CDAI < 200 at 1 week prior to the visit. At Key Visits 3, 4, and 5 (every 12 weeks after Key visit 1), the criteria for a change in treatment were a CDAI decrease of ≥ 100 (CR-100) compared to Baseline or CDAI < 200, and absence of prednisone during the preceding week.
  Interventions: Biological: Adalimumab; Drug: Prednisone; Drug: Azathioprine

INTERVENTIONS:
Biological: Adalimumab — If adalimumab was initiated, it was administered subcutaneously as a 160 mg induction dose the first week, followed by 80 mg 2 weeks later, followed by 40 mg every other week as a maintenance dose. The dose of adalimumab was increased from 40 mg eow to 40 mg every week in participants with an inadequate response and de-escalated to 40 mg eow in participants who met success criteria.
  Other Names: ABT-D2E7; Humira
Drug: Prednisone — The suggested regimen for participants initiating prednisone consisted of a maximum dose of prednisone 40 mg/day for 2 weeks, followed by a fixed taper for 6 weeks.
Drug: Azathioprine — Participants with normal thiopurine methyltransferase (TPMT) enzyme activity could receive oral azathioprine 2.5 mg/kg/day. In participants with intermediate TPMT enzyme activity azathioprine was initiated at a dose of 1.25 mg/kg/day. The dose of azathioprine was adjusted according to abnormalities of white blood cell (WBC) count, platelet count, liver function tests (LFTs; i.e. alanine transaminase [ALT], aspartate transaminase [AST], alkaline phosphatase), lipase, blood urea nitrogen (BUN), and serum creatinine.

SUMMARY:
The primary objective of this study was to demonstrate that tight control of disease activity, using stringent criteria based on Crohn's disease activity Index (CDAI), biomarkers (high sensitivity C-reactive protein [hs-CRP] and fecal calprotectin), and corticosteroid use, improves the rate of mucosal healing 48 weeks after randomization compared with management using less stringent criteria based only on CDAI and corticosteroid use.

DETAILED DESCRIPTION:
The study included a 1- to 3-week screening period, up to 8 weeks of prednisone run-in treatment, a 48-week post-randomization treatment period, and a 70 day follow-up phone call or clinic visit, for a total duration of up to 69 weeks.

Participants who met entry criteria were enrolled and initiated an oral prednisone regimen at Baseline (Week 0). At the first key visit, participants were randomized into 1 of 2 groups (Tight Control group or Clinically Driven group), with stratification according to screening smoking status, weight, and disease duration.

The first key visit was the randomization visit; subsequent key visits occurred every 12 weeks following the first key visit. Randomization normally took place 9 weeks after Baseline. However, participants who fulfilled the early randomization criteria may have been randomized as early as the Baseline (Week 0) visit. Therapeutic option changes, if appropriate, occurred at key visits based on results from previous success criteria visits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ileal, colonic (including rectal), or ileocolonic Crohn's disease (CD) confirmed using imaging technology or endoscopy not more than 6 years prior to Baseline.
* CDAI score of greater than or equal to 220 and less than or equal to 450 at the Baseline visit in participants not receiving prednisone or equivalent at Baseline. CDAI score of greater than or equal to 200 and less than or equal to 450 at the Baseline visit if the participant is receiving prednisone less than or equal to 20 mg or equivalent for at least 7 days before Baseline. CDAI score of greater than 150 and less than or equal to 450 at the Baseline visit if the participant is receiving prednisone higher than 20 mg or equivalent for greater than or equal to 7 days before Baseline
* Participant or his/her legal representative have voluntarily signed and dated an informed consent approved by and compliant with the requirements of this study protocol which has been approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
* Adequate cardiac, renal and hepatic function as determined by the Principal Investigator and demonstrated by Screening laboratory evaluations, questionnaires and physical examination results that do not indicate an abnormal clinical condition which would place the participant at undue risk and thus preclude participation in the study.
* Participant must be able to self-inject and orally administer study medication or have a designee or Healthcare Professional who can assist

Exclusion Criteria:

* Previous or current biologic use for Crohn's disease or participation in a biologic study
* Previous or current use of immunomodulators (e.g., methotrexate, azathioprine, 6-mercaptopurine, JAK inhibitor, alpha-integrin) for Crohn's disease or participation in a Crohn's disease study with immunomodulator(s). Current use of immunomodulators for non-Crohn's disease at Baseline.
* Greater than two previous courses of corticosteroid (systemic corticosteroid) or budesonide) for Crohn's Disease. A course is defined as 1) total duration for burst and taper ≥ 4 weeks and 2) prednisone or equivalent ≥ 40 mg (or budesonide ≥ 9 mg) for at least 2 weeks.
* Participants with a poorly controlled medical condition such as: uncontrolled diabetes with documented history of recurrent infections, unstable ischemic heart disease, moderate to severe congestive heart failure (New York Heart Association [NYHA] class III or IV), recent cerebrovascular accident and any other condition which, in the opinion of the Investigator or the sponsor, would put the participant at risk by participation in the protocol
* Participants with positive C. difficile stool assay at Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2011-02-11 (Actual); Primary Completion 2016-11-03 (Actual); Study Completion 2017-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Robinson, Pharm.D., Study Director — AbbVie

REFERENCES:
- [Derived] Lakatos PL, Kaplan GG, Bressler B, Khanna R, Targownik L, Jones J, Rahal Y, McHugh K, Panaccione R. Cost-Effectiveness of Tight Control for Crohn's Disease With Adalimumab-Based Treatment: Economic Evaluation of the CALM Trial From a Canadian Perspective. J Can Assoc Gastroenterol. 2022 Mar 10;5(4):169-176. doi: 10.1093/jcag/gwac001. eCollection 2022 Aug. PMID 35919766
- [Derived] Ungaro RC, Yzet C, Bossuyt P, Baert FJ, Vanasek T, D'Haens GR, Joustra VW, Panaccione R, Novacek G, Reinisch W, Armuzzi A, Golovchenko O, Prymak O, Goldis A, Travis SP, Hebuterne X, Ferrante M, Rogler G, Fumery M, Danese S, Rydzewska G, Pariente B, Hertervig E, Stanciu C, Serrero M, Diculescu M, Peyrin-Biroulet L, Laharie D, Wright JP, Gomollon F, Gubonina I, Schreiber S, Motoya S, Hellstrom PM, Halfvarson J, Butler JW, Petersson J, Petralia F, Colombel JF. Deep Remission at 1 Year Prevents Progression of Early Crohn's Disease. Gastroenterology. 2020 Jul;159(1):139-147. doi: 10.1053/j.gastro.2020.03.039. Epub 2020 Mar 26. PMID 32224129
- [Derived] Panaccione R, Colombel JF, Travis SPL, Bossuyt P, Baert F, Vanasek T, Danalioglu A, Novacek G, Armuzzi A, Reinisch W, Johnson S, Buessing M, Neimark E, Petersson J, Lee WJ, D'Haens GR. Tight control for Crohn's disease with adalimumab-based treatment is cost-effective: an economic assessment of the CALM trial. Gut. 2020 Apr;69(4):658-664. doi: 10.1136/gutjnl-2019-318256. Epub 2019 Jul 8. PMID 31285357
- [Derived] Colombel JF, Panaccione R, Bossuyt P, Lukas M, Baert F, Vanasek T, Danalioglu A, Novacek G, Armuzzi A, Hebuterne X, Travis S, Danese S, Reinisch W, Sandborn WJ, Rutgeerts P, Hommes D, Schreiber S, Neimark E, Huang B, Zhou Q, Mendez P, Petersson J, Wallace K, Robinson AM, Thakkar RB, D'Haens G. Effect of tight control management on Crohn's disease (CALM): a multicentre, randomised, controlled phase 3 trial. Lancet. 2017 Dec 23;390(10114):2779-2789. doi: 10.1016/S0140-6736(17)32641-7. Epub 2017 Oct 31. PMID 29096949
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 59 sites in Canada, European Union, Israel, Japan, Russia, South Africa, Switzerland, Turkey, and the Ukraine.
  The study included a screening period, up to 8 weeks of prednisone run-in treatment, a 48-week post-randomization treatment period, and a 70 day follow-up phone call or clinic visit.
Pre-assignment Details: A total of 252 participants were enrolled and received study treatment, of whom
  * 165 entered the prednisone run-in
    * 157 randomized (45 prior to Week 9, 112 at Week 9)
    * 8 discontinued prior to randomization.
  * 87 randomized at Baseline.
  Randomization was stratified by smoking status, weight, and disease duration.
Period: Overall Study
Arm/Group | Clinically Driven Management | Tight Control Management
Started | 122 (Total randomized includes participants who randomized at Week 9 and earlier.) | 122 (Total randomized includes participants who randomized at Week 9 and earlier.)
Early Randomized (Baseline to Week 9) | 63 | 69
Randomized at Week 9 | 59 | 53
Completed | 93 | 90
Not Completed | 29 | 32
Not completed — Adverse Event | 12 | 16
Not completed — Lack of Efficacy | 12 | 5
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Miscellaneous | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Clinically Driven Management: Participants randomized to receive management of disease activity using criteria based on Crohn's Disease Activity Index (CDAI) and corticosteroid use.
  Participants received customized therapy that could include prednisone, adalimumab, and azathioprine.
- Tight Control Management: Participants randomized to receive management of disease activity using criteria based on Crohn's Disease Activity Index (CDAI), high sensitivity C-reactive protein (hs-CRP), fecal calprotectin, and corticosteroid use.
  Participants received customized therapy that could include prednisone, adalimumab, and azathioprine.
- Total: Total of all reporting groups
Arm/Group | Clinically Driven Management | Tight Control Management | Total
Number analyzed (Participants) | 122 | 122 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.10 (11.40) | 32.10 (11.97) | 31.60 (11.67)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 97 | 96 | 193
  40 to < 65 years | 23 | 24 | 47
  ≥ 65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 72 | 141
  Male | 53 | 50 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 113 | 113 | 226
  Black | 2 | 3 | 5
  Asian | 3 | 2 | 5
  American Indian/Alaska Native | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Multi-race | 1 | 1 | 2
  Other | 3 | 3 | 6
Weight [Count of Participants; unit: Participants]
  < 70 kg | 79 | 81 | 160
  ≥ 70 kg | 43 | 41 | 84
Current Tobacco Use [Count of Participants; unit: Participants]
  Yes | 33 | 31 | 64
  No | 89 | 91 | 180
Disease Duration [Count of Participants; unit: Participants]
  ≤ 2 years | 106 | 106 | 212
  > 2 years | 16 | 16 | 32
Crohn's Disease Endoscopy Index of Severity (CDEIS) [Mean (Standard Deviation); unit: units on a scale] — CDEIS is an index for determining the severity of Crohn's disease. The CDEIS considers deep ulcerations, superficial ulcerations, ulcerated and non-ulcerated surface, and the presence of ulcerated/non-ulcerated stenosis evaluated in 5 pre-defined segments of the colon (ileum, ascending colon, transverse colon, descending colon and sigmoid loop, and rectum). The score ranges from 0 to 44 where higher scores indicate more severe endoscopic activity.
  units on a scale | 14.26 (6.925) | 13.38 (6.049) | 13.82 (6.503)
Crohn's Disease Activity Index (CDAI) [Mean (Standard Deviation); unit: units on a scale] — CDAI is a tool used to quantify the symptoms of patients with Crohn's disease. Participants were asked to record the frequency of stools, abdominal pain and general well-being on a daily basis. In addition to the diary data, the investigator assessed the following for the calculation of CDAI: presence of complications, the use of antidiarrheal medicines, presence of an abdominal mass, hematocrit, and body weight. The CDAI is the sum of the products of each item multiplied by a weighting factor and generally ranges from 0 up to 600, where higher scores indicate more severe disease.
  units on a scale | 267.7 (58.35) | 273.3 (59.48) | 270.5 (58.86)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Mucosal Healing and No Deep Ulcerations
Description: Percentage of participants with mucosal healing (defined as Crohn's disease endoscopy Index of severity [CDEIS] < 4) and no deep ulcerations on ileocolonoscopy (defined as the absence of all deep ulcerations in all segments explored in CDEIS) at 48 weeks after randomization (48 weeks after the 1st Key visit). The ileocolonoscopies were evaluated by the site.
  CDEIS is an index for determining the severity of Crohn's disease. The CDEIS considers deep ulcerations, superficial ulcerations, ulcerated and non-ulcerated surface, and the presence of ulcerated/non-ulcerated stenosis evaluated in 5 pre-defined segments of the colon (ileum, ascending colon, transverse colon, descending colon and sigmoid loop, and rectum). The score ranges from 0 to 44 where higher scores indicate more severe endoscopic activity.
  Participants with missing data 48 weeks after Randomization were counted as non-responders.
Time Frame: 48 weeks after Randomization
Population: All randomized participants; Participants with missing CDEIS values from endoscopies performed 48 weeks after randomization were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
percentage of participants | 30.3 | 45.9
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.010, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test stratified by Screening smoking status (yes or no) and weight (< 70 kg or ≥ 70 kg)

2. Secondary Outcome: Percentage of Participants in Deep Remission 48 Weeks After Randomization
Description: Deep remission was defined as CDAI < 150, discontinuation from steroids for at least 8 weeks, absence of draining fistula, CDEIS < 4 and no deep ulcerations.
  CDAI is a tool used to quantify the symptoms of patients with Crohn's disease. The score includes the frequency of stools, abdominal pain and general well-being as well as the presence of complications, use of antidiarrheals, presence of abdominal mass, hematocrit and weight. CDAI generally ranges from 0 to 600 where higher scores indicate more severe disease.
  CDEIS is an index for determining the severity of Crohn's disease. The CDEIS considers deep ulcerations, superficial ulcerations, ulcerated and non-ulcerated surface, and the presence of ulcerated/non-ulcerated stenosis evaluated in 5 pre-defined segments of the colon. The range of the score is from 0 to 44 where higher scores indicate more severe endoscopic activity.
  Participants with missing data 48 weeks after randomization were counted as non-responders.
Time Frame: 48 weeks after Randomization
Population: All randomized participants; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
percentage of participants | 23.0 | 36.9
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.014, Cochran-Mantel-Haenszel; CMH test stratified by screening smoking status (yes or no) and weight (< 70 kg, ≥ 70 kg)

3. Secondary Outcome: Percentage of Participants in Biologic Remission 48 Weeks After Randomization
Description: Biologic remission was defined as high sensitivity C-reactive protein (hs-CRP) < 5 mg/L, fecal Calprotectin < 250 μg/g, and CDEIS < 4 at 48 weeks after randomization.
  CDEIS is an index for determining the severity of Crohn's disease. The CDEIS considers deep ulcerations, superficial ulcerations, ulcerated and non-ulcerated surface, and the presence of ulcerated/non-ulcerated stenosis evaluated in 5 pre-defined segments of the colon. The range of the score is from 0 to 44 where higher scores indicate more severe endoscopic activity.
  Participants with missing values 48 weeks after Randomization were counted as non-responders.
Time Frame: 48 weeks after Randomization
Population: All randomized participants; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
percentage of participants | 15.6 | 29.5
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel; CMH test stratified by screening smoking status (yes or no) and weight (< 70 kg, ≥ 70 kg)

4. Secondary Outcome: Percentage of Participants With Mucosal Healing 48 Weeks After Randomization
Description: Percentage of participants with mucosal healing (defined as a CDEIS < 4) at 48 weeks after randomization (48 weeks after the 1st Key visit). The ileocolonoscopies were evaluated by the site.
  CDEIS is an index for determining the severity of Crohn's disease. The CDEIS considers deep ulcerations, superficial ulcerations, ulcerated and non-ulcerated surface, and the presence of ulcerated/non-ulcerated stenosis evaluated in 5 pre-defined segments of the colon. The range of the score is from 0 to 44 where higher scores indicate more severe endoscopic activity.
  Participants with missing values 48 weeks after Randomization were counted as non-responders.
Time Frame: 48 weeks after Randomization
Population: All randomized participants; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
percentage of participants | 30.3 | 45.9
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.010, Cochran-Mantel-Haenszel; CMH test stratified by screening smoking status (yes or no) and weight (< 70 kg, ≥ 70 kg)

5. Secondary Outcome: Percentage of Participants With Mucosal Healing and CDEIS < 4 in Every Segment 48 Weeks After Randomization
Description: Percentage of participants with mucosal healing (defined as CDEIS < 4) and CDEIS < 4 in every segment on ileocolonoscopy at 48 weeks after randomization. The ileocolonoscopies were evaluated by the site.
  CDEIS is an index for determining the severity of Crohn's disease. The CDEIS considers deep ulcerations, superficial ulcerations, ulcerated and non-ulcerated surface, and the presence of ulcerated/non-ulcerated stenosis evaluated in 5 pre-defined segments of the colon. The range of the score is from 0 to 44 where higher scores indicate more severe endoscopic activity.
  Participants with missing values 48 weeks after randomization were counted as non-responders.
Time Frame: 48 weeks after Randomization
Population: All randomized participants; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
percentage of participants | 23.8 | 29.5
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.299, Cochran-Mantel-Haenszel; CMH test stratified by screening smoking status (yes or no) and weight (< 70 kg, ≥ 70 kg)

6. Secondary Outcome: Percentage of Participants With Complete Mucosal Healing 48 Weeks After Randomization
Description: Complete mucosal healing was defined as CDEIS = 0. CDEIS is an index for determining the severity of Crohn's disease. The CDEIS considers deep ulcerations, superficial ulcerations, ulcerated and non-ulcerated surface, and the presence of ulcerated/non-ulcerated stenosis evaluated in 5 pre-defined segments of the colon. The range of the score is from 0 to 44 where higher scores indicate more severe endoscopic activity.
  Participants with missing values 48 weeks after randomization were counted as non-responders.
Time Frame: 48 weeks after Randomization
Population: All randomized participants; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
percentage of participants | 16.4 | 18.0
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.728, Cochran-Mantel-Haenszel; CMH test stratified by screening smoking status (yes or no) and weight (< 70 kg, ≥ 70 kg)

7. Secondary Outcome: Percentage of Participants With Endoscopic Response 48 Weeks After Randomization
Description: Endoscopic response was defined as a decrease CDEIS > 5 points. CDEIS is an index for determining the severity of Crohn's disease. The CDEIS considers deep ulcerations, superficial ulcerations, ulcerated and non-ulcerated surface, and the presence of ulcerated/non-ulcerated stenosis evaluated in 5 pre-defined segments of the colon. The range of the score is from 0 to 44 where higher scores indicate more severe endoscopic activity.
  Participants with missing values 48 weeks after Randomization were counted as non-responders.
Time Frame: 48 weeks after Randomization
Population: All randomized participants; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
percentage of participants | 40.2 | 50.8
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.067, Cochran-Mantel-Haenszel; CMH test stratified by screening smoking status (yes or no) and weight (< 70 kg, ≥ 70 kg)

8. Secondary Outcome: Change From Baseline in CDEIS at 48 Weeks After Randomization
Description: CDEIS is an index for determining the severity of Crohn's disease. The CDEIS considers deep ulcerations, superficial ulcerations, ulcerated and non-ulcerated surface, and the presence of ulcerated/non-ulcerated stenosis evaluated in 5 pre-defined segments of the colon (ileum, ascending colon, transverse colon, descending colon and sigmoid loop, and rectum). The score ranges from 0 to 44 where higher scores indicate more severe endoscopic activity. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 48 weeks after Randomization
Population: Randomized participants with non-missing data at Baseline and 48 weeks after Randomization.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 96 | 105
units on a scale | -6.4 (7.69) | -7.7 (7.25)
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.116, ANCOVA; Model included factors for treatment group, screening smoking status (yes or no), and weight (< 70 kg, ≥ 70 kg), and Baseline values as covariate; LS Mean Difference = -1.4, 95% CI 2-sided [-3.2 to 0.4]

9. Secondary Outcome: Change From Baseline in CDAI Over Time
Description: The Crohn's Disease Activity Index (CDAI) is a research tool used to quantify the symptoms of patients with Crohn's disease. Participants were asked to record the frequency of stools, abdominal pain and general well-being on a daily basis. In addition to the diary data, the investigator assessed the following for the calculation of CDAI: presence of complications (arthritis/arthralgia, iritis/uveitis, erythema nodosum/pyoderma gangrenosum/aphthous stomatitis, anal fissure/fistula/abscess, other fistula, and fever), the use of antidiarrheal medicines, presence of an abdominal mass, hematocrit, and body weight. The CDAI is the sum of the products of each item multiplied by a weighting factor and generally ranges from 0 up to 600, where remission of Crohn's disease is defined as CDAI < 150, and severe disease is defined as CDAI > 450. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 4 and 8 weeks during the prednisone run-in, and 2, 6, 11, 14, 18, 23, 26, 30, 35, 38, 42, and 48 weeks after Randomization.
Population: Randomized participants with non-missing data at each time point. CDAI was only measured at 14, 18, 26, 30, 38 and 42 weeks after randomization if a participant had initiated a change in treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
units on a scale
  Week 4 of Prednisone Run-in: number analyzed (Participants) | 79 | 76
  Week 4 of Prednisone Run-in | -78.3 (80.02) | -90.9 (81.53)
  Week 8 of Prednisone Run-in: number analyzed (Participants) | 62 | 54
  Week 8 of Prednisone Run-in | -64.2 (90.48) | -105.5 (88.40)
  2 Weeks After Randomization: number analyzed (Participants) | 95 | 110
  2 Weeks After Randomization | -80.2 (82.27) | -110.1 (85.06)
  6 Weeks After Randomization: number analyzed (Participants) | 100 | 110
  6 Weeks After Randomization | -93.1 (100.81) | -130.8 (89.40)
  11 Weeks After Randomization: number analyzed (Participants) | 114 | 115
  11 Weeks After Randomization | -103.5 (98.65) | -141.0 (97.82)
  14 Weeks After Randomization: number analyzed (Participants) | 26 | 16
  14 Weeks After Randomization | -71.1 (89.18) | -101.2 (115.90)
  18 Weeks After Randomization: number analyzed (Participants) | 27 | 16
  18 Weeks After Randomization | -69.9 (78.95) | -112.0 (115.01)
  23 Weeks After Randomization: number analyzed (Participants) | 97 | 107
  23 Weeks After Randomization | -143.3 (97.83) | -154.1 (101.63)
  26 Weeks After Randomization: number analyzed (Participants) | 20 | 42
  26 Weeks After Randomization | -71.8 (129.09) | -135.7 (112.43)
  30 Weeks After Randomization: number analyzed (Participants) | 20 | 42
  30 Weeks After Randomization | -47.9 (143.75) | -143.8 (103.54)
  35 Weeks After Randomization: number analyzed (Participants) | 92 | 95
  35 Weeks After Randomization | -140.4 (104.83) | -166.4 (93.12)
  38 Weeks After Randomization: number analyzed (Participants) | 15 | 19
  38 Weeks After Randomization | -60.8 (83.51) | -132.8 (103.15)
  42 Weeks After Randomization: number analyzed (Participants) | 11 | 16
  42 Weeks After Randomization | -76.8 (78.53) | -107.4 (99.19)
  48 Weeks After Randomization: number analyzed (Participants) | 82 | 90
  48 Weeks After Randomization | -146.2 (102.87) | -175.8 (97.69)

10. Secondary Outcome: Time to Crohn's Disease Flare
Description: Time to Crohn's disease flare, where flare is defined as an increase in CDAI ≥ 70 points compared to Week 8 or Early Randomization CDAI, and a CDAI > 220.
Time Frame: From Randomization to 48 weeks after Randomization
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
days | NA [NA to NA] — Could not be estimated due to the low number of flare events | NA [NA to NA] — Could not be estimated due to the low number of flare events
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.012, Regression, Cox; Cox Proportional Hazard = 0.442, 95% CI 2-sided [0.2 to 0.8]

11. Secondary Outcome: Time to Clinical Remission
Description: Clinical remission was defined as CDAI < 150. CDAI is a tool used to quantify the symptoms of patients with Crohn's disease. The score includes the frequency of stools, abdominal pain and general well-being as well as the presence of complications, use of antidiarrheals, presence of abdominal mass, hematocrit and weight. CDAI scores generally range from 0 to 600 where higher scores indicate more severe disease.
Time Frame: From Randomization through 48 weeks after Randomization
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
days | 78 [28 to 163] | 43 [15 to 101]
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.008, Regression, Cox; Cox Proportional Hazard = 1.450, 95% CI 2-sided [1.1 to 1.9]

12. Secondary Outcome: Time to Steroid-free Remission
Description: Steroid-free remission was defined as CDAI < 150 and discontinuation from steroids for at least 8 weeks. CDAI is a tool used to quantify the symptoms of patients with Crohn's disease. The score includes the frequency of stools, abdominal pain and general well-being as well as the presence of complications, use of antidiarrheals, presence of abdominal mass, hematocrit and weight. CDAI generally ranges from 0 to 600 where higher scores indicate more severe disease.
Time Frame: From Randomization through 48 weeks after Randomization
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
days | 162 [80 to 255] | 159 [78 to 168]
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.052, Regression, Cox; Cox Proportional Hazard = 1.337, 95% CI 2-sided [1.0 to 1.8]

13. Secondary Outcome: Percentage of Participants in Clinical Remission Over Time
Description: Clinical remission was defined as CDAI < 150. CDAI is a tool used to quantify the symptoms of patients with Crohn's disease. The score includes the frequency of stools, abdominal pain and general well-being as well as the presence of complications, use of antidiarrheals, presence of abdominal mass, hematocrit and weight. CDAI generally ranges from 0 to 600 where higher scores indicate more severe disease.
  Participants with missing data at each time point were counted as non-responders.
Time Frame: as for outcome 9
Population: Randomized participants; non-responder imputation was used. CDAI was only measured at 14, 18, 26, 30, 38 and 42 weeks after randomization if a participant had initiated a change in treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
percentage of participants
  Week 4 of Prednisone Run-in | 24.6 | 30.3
  Week 8 of Prednisone Run-in | 14.8 | 22.1
  2 Weeks After Randomization | 23.8 | 41.0
  6 Weeks After Randomization | 32.8 | 47.5
  11 Weeks After Randomization | 41.8 | 62.3
  14 Weeks After Randomization | 8.2 | 6.6
  18 Weeks After Randomization | 9.0 | 8.2
  23 Weeks After Randomization | 50.8 | 65.6
  26 Weeks After Randomization | 4.1 | 20.5
  30 Weeks After Randomization | 3.3 | 23.0
  35 Weeks After Randomization | 45.1 | 59.8
  38 Weeks After Randomization | 4.1 | 9.0
  42 Weeks After Randomization | 4.1 | 7.4
  48 Weeks After Randomization | 43.4 | 59.8

14. Secondary Outcome: Percentage of Participants in Steroid-free Remission Over Time
Description: Steroid-free remission was defined as CDAI < 150 and discontinuation from steroids for at least 8 weeks. CDAI is a tool used to quantify the symptoms of patients with Crohn's disease. The score includes the frequency of stools, abdominal pain and general well-being as well as the presence of complications, use of antidiarrheals, presence of abdominal mass, hematocrit and weight. CDAI generally ranges from 0 to 600 where higher scores indicate more severe disease.
  Participants with missing data at each time point were counted as non-responders.
Time Frame: 11, 14, 18, 23, 26, 30, 35, 38, 42, and 48 weeks after Randomization.
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
percentage of participants
  11 Weeks After Randomization | 23.8 | 39.3
  14 Weeks After Randomization | 4.1 | 4.9
  18 Weeks After Randomization | 3.3 | 7.4
  23 Weeks After Randomization | 45.1 | 63.1
  26 Weeks After Randomization | 2.5 | 18.9
  30 Weeks After Randomization | 0.8 | 21.3
  35 Weeks After Randomization | 42.6 | 59.0
  38 Weeks After Randomization | 4.1 | 9.0
  42 Weeks After Randomization | 4.1 | 7.4
  48 Weeks After Randomization | 39.3 | 59.8

15. Secondary Outcome: Time to All-cause Hospitalization
Description: Hospitalization was defined as a visit to hospital/clinic resulting in admission and overnight stay in hospital/clinic.
Time Frame: From Randomization through 48 weeks after Randomization
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
days | NA [NA to NA] — Could not be estimated due to the low number of hospitalization events | NA [NA to NA] — Could not be estimated due to the low number of hospitalization events
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.501, Regression, Cox; Cox Proportional Hazard = 0.823, 95% CI 2-sided [0.5 to 1.5]

16. Secondary Outcome: Time to Crohn's Disease-related Hospitalization or Hospitalization Due to Adverse Event Relating to Study Medication
Description: Crohn's disease-related hospitalization was defined as a visit to hospital/clinic resulting in admission and overnight stay in hospital/clinic for reasons related to Crohn's disease (CD). Hospitalization for adverse events relating to study medication, i.e., prednisone, azathioprine or adalimumab, were according to Investigator's clinical judgment.
Time Frame: From Randomization through 48 weeks after Randomization
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
days | NA [NA to NA] — Could not be estimated due to the low number of hospitalization events | NA [NA to NA] — Could not be estimated due to the low number of hospitalization events
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.459, Regression, Cox; Cox Proportional Hazard = 0.785, 95% CI 2-sided [0.4 to 1.5]

17. Secondary Outcome: Number of Major Crohn's Disease-related Surgeries After Randomization
Description: Major Crohn's disease-related intra-abdominal surgery included:
  * bowel resection
  * ostomy
  * by-pass
  * strictureplasty
  * drainage of abdominal or pelvic abscess (surgical drainage or percutaneous drainage by interventional radiology).
  The following were excluded:
  * debridement
  * exploration laparotomy
  * abdominal surgery for other reason
  * perineal related surgery
  * abscess drainage
  * placement of setons
  * fistulotomy
  * Total parental nutrition (TPN) use
Time Frame: From Randomization through 48 weeks after Randomization
Population: All randomized participants
Measure: Number; unit: surgeries
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
surgeries | 3 | 6

18. Secondary Outcome: Number of Crohn's Disease-related Hospitalizations After Randomization
Description: Any hospitalization with an overnight stay in hospital/clinic related to Crohn's disease.
Time Frame: From Randomization through 48 weeks after Randomization
Population: All randomized participants
Measure: Number; unit: hospitalizations
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
hospitalizations | 29 | 14

19. Secondary Outcome: Number of All-cause Hospitalizations After Randomization
Description: Hospitalization was defined as a visit to hospital/clinic resulting in admission and overnight stay in hospital/clinic.
Time Frame: From Randomization through 48 weeks after Randomization
Population: All randomized participants
Measure: Number; unit: hospitalizations
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
hospitalizations | 37 | 25

20. Secondary Outcome: Total Length of Stay in Hospital for All-cause Hospitalizations
Time Frame: From Randomization through 48 weeks after Randomization
Population: Randomized participants with all-cause hospitalizations
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 26 | 22
days | 40.2 (45.72) | 50.1 (85.69)

21. Secondary Outcome: Total Length of Stay in Hospital for Crohn's Disease-related Hospitalizations
Time Frame: From Randomization through 48 weeks after Randomization
Population: Randomized participants with Crohn's disease-related hospitalizations
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 21 | 13
days | 9.8 (7.21) | 15.8 (20.39)

22. Secondary Outcome: Number of Crohn's Disease-related Surgical Procedures After Randomization
Description: The total number of CD-related surgical procedures included major CD-related surgery, debridement, perineal related surgery - abscess drainage, seton placement, fistulotomy, and TPN.
Time Frame: From Randomization through 48 weeks after Randomization
Population: All randomized participants
Measure: Number; unit: surgical procedures
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
surgical procedures | 9 | 7

23. Secondary Outcome: Time to Crohn's Disease-related Hospitalization Due to Emergency
Description: Hospitalization was defined as a visit to hospital/clinic resulting in admission and overnight stay in hospital/clinic. Hospitalization due to emergency was defined as a hospitalization admitted through the emergency department.
Time Frame: From Randomization through 48 weeks after Randomization
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
days | NA [NA to NA] — Could not be estimated due to the low number of emergency hospitalizations | NA [NA to NA] — Could not be estimated due to the low number of emergency hospitalizations
Statistical Analysis 1: Comparison: Clinically Driven Management vs Tight Control Management; Test type: Superiority; p = 0.212, Regression, Cox; Cox Proportional Hazard = 0.423, 95% CI 2-sided [0.1 to 1.6]

24. Secondary Outcome: Number of Crohn's Disease-related Hospitalizations Due to Emergency
Description: as for outcome 23
Time Frame: From Randomization through 48 weeks after Randomization
Population: All randomized participants
Measure: Number; unit: emergency hospitalizations
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
emergency hospitalizations | 11 | 4

25. Secondary Outcome: Change in Crohn's Disease Behavior According to Montreal Classification
Description: Participants' Crohn's Disease was classified according to the Montreal Classification which classifies CD according to its predominant phenotypic elements (age at diagnosis, location, and disease behavior) based on the results of clinical examination and endoscopy.
  Disease behavior was classified according to the following:
  B1 = non-stricturing, non-penetrating; B2 = structuring; B3 = penetrating; P = perianal disease modifier.
  The change in Montreal Classification is presented in three categories: no change, deterioration, and improvement. Deterioration was defined as an increase in behavior index between 1 and 3, or development of perianal disease. Participants with missing data at Week 48 were classified as deterioration.
Time Frame: From Baseline to 48 weeks after Randomization
Population: All randomized participants; non-responder imputation was used.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
Participants
  Deterioration | 54 | 35
  No Change | 64 | 79
  Improvement | 4 | 8

26. Secondary Outcome: Change From Baseline in High Sensitivity C-Reactive Protein (Hs-CRP) Over Time
Description: High sensitivity C-reactive protein was analyzed by a central laboratory.
Time Frame: Baseline and 8 weeks during the prednisone run-in, and 11, 23, 35, and 48 weeks after Randomization.
Population: Randomized participants; last observation carried forward imputation was used.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 122
mg/L
  Week 8 of Prednisone Run-in: number analyzed (Participants) | 77 | 73
  Week 8 of Prednisone Run-in | -10.3 (40.04) | -9.2 (33.67)
  11 Weeks After Randomization: number analyzed (Participants) | 120 | 121
  11 Weeks After Randomization | -14.6 (31.87) | -15.9 (26.38)
  23 Weeks After Randomization: number analyzed (Participants) | 121 | 122
  23 Weeks After Randomization | -15.1 (31.59) | -14.7 (28.94)
  35 Weeks After Randomization: number analyzed (Participants) | 121 | 122
  35 Weeks After Randomization | -11.0 (31.22) | -14.0 (28.85)
  48 Weeks After Randomization: number analyzed (Participants) | 121 | 122
  48 Weeks After Randomization | -12.3 (28.97) | -13.2 (28.93)

27. Secondary Outcome: Change in Fecal Calprotectin From Baseline to 48 Weeks After Randomization
Description: Stool samples were analyzed by a central laboratory for fecal calprotectin qualitative measurement (< 250 or ≥ 250 μg/g). Results are reported for participants in each category at Baseline and 48 weeks after Randomization.
  Participants with missing data 48 weeks after Randomization were counted as having fecal calprotectin ≥ 250µg/g.
Time Frame: Baseline and 48 weeks after Randomization
Population: Randomized participants with Baseline data; non-responder imputation was used.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 122 | 120
Participants
  Baseline < 250µg/g and Week 48 < 250µg/g | 8 | 14
  Baseline < 250µg/g and Week 48 ≥ 250µg/g | 9 | 10
  Baseline ≥ 250µg/g and Week 48 < 250µg/g | 37 | 44
  Baseline ≥ 250µg/g and Week 48 ≥ 250µg/g | 68 | 52

28. Secondary Outcome: Total Dose of Prednisone
Description: The total dose of prednisone each participant received during both the run-in phase and post-randomization treatment phase.
Time Frame: From Baseline through 48 weeks after Randomization
Population: Participants who received prednisone
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 102 | 104
mg | 1505.7 (1029.83) | 1369.8 (1137.65)

29. Secondary Outcome: Change From Baseline in Quality of Life in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score
Description: The IBDQ measures the effects of inflammatory bowel disease on daily function and quality of life. The IBDQ consists of 32 questions which address symptoms as a result of Crohn's disease, feeling in general, and mood. Each question is answered on a scale from 1 (all of the time) to 7 ( none of the time); the total score ranges from 7 (worst) to 224 (best). A positive change from baseline indicates improvement.
Time Frame: Baseline and 48 weeks after Randomization
Population: Randomized participants with baseline and at least one post-baseline value; last observation carried forward imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 111 | 111
units on a scale | 31.2 (39.33) | 41.9 (36.90)

30. Secondary Outcome: Change From Baseline in Work Productivity Activity Index - Crohn's Disease (WPAI:CD)
Description: The WPAI:CD questionnaire was used to assess impairments in both paid work and unpaid work due to symptoms of Crohn's Disease. The self-administered questionnaire consisted of 6 questions.
  Work time missed was defined as the percentage of time absent from work due to Crohn's disease in the past week.
  Impairment while working is the participant's assessment of the degree to which Crohn's disease affected productivity while working in the past 7 days.
  Total work productivity impairment takes into account both hours missed due to Crohn's disease symptoms and the patient's assessment of the degree to which Crohn's disease affected their productivity while working.
  Total activity impairment is the percent impairment of non-work related activities due to Crohn's disease.
  WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 48 weeks after Randomization
Population: Randomized participants with baseline and at least one post-baseline value; last observation carried forward imputation was used. The first 3 scores were only calculated for participants who were employed.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 119 | 118
percent impairment
  Work time missed: number analyzed (Participants) | 67 | 62
  Work time missed | -12.8 (30.17) | -17.6 (41.33)
  Impairment while working: number analyzed (Participants) | 64 | 52
  Impairment while working | -17.5 (23.37) | -25.8 (34.32)
  Overall work impairment: number analyzed (Participants) | 67 | 62
  Overall work impairment | -21.7 (29.68) | -29.2 (39.53)
  Activity impairment: number analyzed (Participants) | 118 | 118
  Activity impairment | -19.2 (27.16) | -27.7 (33.22)

31. Secondary Outcome: Change From Baseline in Patient Health Questionnaire - 9 (PHQ9)
Description: The PHQ-9 is a 9-item questionnaire for assessing the severity of depression. Each question is answered on a scale from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27, where higher scores indicate more severe depression. A negative change from Baseline score indicates improvement.
Time Frame: Baseline and 48 weeks after Randomization
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 120 | 120
units on a scale | -3.6 (5.65) | -5.6 (5.95)

32. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score
Description: The FACIT-Fatigue scale is a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, from 0 (not at all) to 4 (very much). The FACIT-Fatigue score ranges from 0 to 52, with higher scores denoting lower levels of fatigue.
  A positive change from Baseline score indicates an improvement.
  .
Time Frame: Baseline and 48 weeks after Randomization
Population: Randomized participants with Baseline and at least 1 post-baseline value; last observation carried forward imputation was used
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 120 | 119
units on a scale | 7.6 (10.85) | 13.0 (13.19)

33. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Summary and Mental Component Summary Scores
Description: The Medical Outcome Study Short Form 36-Item Health Survey (SF-36), Version 2 is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component summary (PCS) score summarizes the subscales physical functioning, role-physical, bodily pain, and general health. The mental component summary (MCS) score summarizes the subscales vitality, social functioning, role-emotional, and mental health. Each score ranges from 0 to 100 where higher scores indicate a better quality of life. A positive change from Baseline score indicates an improvement.
Time Frame: Baseline and 48 weeks after Randomization
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinically Driven Management | Tight Control Management
Number analyzed (Participants) | 119 | 118
units on a scale
  Physical Component Summary Score | 6.3 (8.34) | 9.2 (10.22)
  Mental Component Summary Score | 5.8 (12.24) | 9.3 (12.40)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from randomization until 70 days after the last dose of study drug (up to 58 weeks).
Description: TEAEs and TESAEs are defined as any adverse event or serious adverse event that begins or worsens in severity on or after randomization until 70 days after the last dose of study drug.
Arm/Group | Clinically Driven Management | Tight Control Management
Serious Adverse Events (participants affected / at risk) | 25/122 | 22/122
Other Adverse Events (participants affected / at risk) | 78/122 | 76/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clinically Driven Management (N=122) | Tight Control Management (N=122)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
ANAL FISTULA (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 12 | 6
ENTERITIS (Gastrointestinal disorders) | 1 | 0
FISTULA OF SMALL INTESTINE (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
ILEAL STENOSIS (Gastrointestinal disorders) | 0 | 2
ILEUS (Gastrointestinal disorders) | 0 | 1
MALOCCLUSION (Gastrointestinal disorders) | 0 | 1
PERITONEAL PERFORATION (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 1
SUBILEUS (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
DRUG INTOLERANCE (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 2
ABSCESS (Infections and infestations) | 1 | 1
ANAL ABSCESS (Infections and infestations) | 4 | 0
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 | 2
ERYSIPELAS (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0
GASTROENTERITIS SALMONELLA (Infections and infestations) | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0
NASAL VESTIBULITIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 | 1
ROTAVIRUS INFECTION (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
VIRAEMIA (Infections and infestations) | 1 | 0
CARTILAGE INJURY (Injury, poisoning and procedural complications) | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 2 | 0
RETROGNATHIA (Musculoskeletal and connective tissue disorders) | 0 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0
CHOLESTEATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 0 | 1
INTRACRANIAL VENOUS SINUS THROMBOSIS (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NASAL SEPTUM DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clinically Driven Management (N=122) | Tight Control Management (N=122)
ANAEMIA (Blood and lymphatic system disorders) | 7 | 8
ABDOMINAL PAIN (Gastrointestinal disorders) | 15 | 13
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 | 8
CROHN'S DISEASE (Gastrointestinal disorders) | 23 | 11
DIARRHOEA (Gastrointestinal disorders) | 2 | 10
NAUSEA (Gastrointestinal disorders) | 7 | 21
VOMITING (Gastrointestinal disorders) | 4 | 13
FATIGUE (General disorders) | 11 | 11
INJECTION SITE ERYTHEMA (General disorders) | 0 | 8
PYREXIA (General disorders) | 12 | 9
INFLUENZA (Infections and infestations) | 8 | 7
NASOPHARYNGITIS (Infections and infestations) | 18 | 18
TONSILLITIS (Infections and infestations) | 1 | 7
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 19 | 17
DIZZINESS (Nervous system disorders) | 7 | 7
HEADACHE (Nervous system disorders) | 15 | 18
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 | 7
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 10 | 4
ALOPECIA (Skin and subcutaneous tissue disorders) | 8 | 5
RASH (Skin and subcutaneous tissue disorders) | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.